CLINICAL TRIAL: NCT07217392
Title: Left Bundle Branch Area Pacing (LBBAP) PMCF Study
Acronym: LBBAP PMCF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10551
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Bradycardia; Right Ventricular Pacing; Heart Failure; Atrial Fibrillation (AF); Cardiac Disease; Left Bundle Branch Area Pacing; Conduction System Pacing
Keywords: Right ventricular pacing; cardiac disease; heart failure; atrial fibrillation; bradycardia; left bundle branch area pacing; conduction system pacing
MeSH Terms: conditions — Bradycardia; Heart Failure; Atrial Fibrillation; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Left Bundle Branch Area Pacing Lead Implant (Experimental): Data will be collected from patients implanted with either the Tendril STS 2088TC or UltiPace LPA1231 lead in the left bundle branch area for pacing and sensing from implant through 6 months. Leads are indicated for use in combination with a compatible pacemaker, implantable cardioverter defibrillator, or cardiac resynchronization therapy device.
  Interventions: Device: LBBAP lead

INTERVENTIONS:
Device: LBBAP lead — The lead is bipolar, steroid-eluting, active fixation, MR Conditional, implantable pacing leads that can be placed in the right atrium, right ventricle, or left bundle branch area for pacing and sensing.
  Other Names: CSP lead

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of LBBA pacing/sensing in patients implanted with the Tendril STS 2088TC or UltiPace LPA1231 lead through 6 months post-implant.

DETAILED DESCRIPTION:
The Left Bundle Branch Area Pacing (LBBAP) Post-Market Clinical Follow-up (PMCF) Study is a global, prospective, single-arm, multi-center trial conducted to support an indication expansion of the Tendril STS (model 2088TC) and UltiPace (model LPA1231) leads to include pacing/sensing in the left bundle branch area (LBBA).

ELIGIBILITY:
Inclusion Criteria:

1. Meets current clinical practice guidelines for implantation of Tendril STS 2088TC or UltiPace LPA1231 lead in the Left Bundle Branch Area
2. Are ≥ 18 years of age or age of legal consent, whichever age is greater.
3. Subject is willing to comply with clinical investigation procedures and agrees to return to clinic for all required follow-up visits, tests, and exams.
4. Subject has been informed of the nature of the clinical investigation, agrees to its provisions and has provided a signed written informed consent, approved by the IRB/EC.

Exclusion Criteria:

1. Patient meets a standard contraindication for lead implant including:

   1. the presence of tricuspid atresia
   2. patients with mechanical tricuspid valves
   3. patients who are expected to be hypersensitive to a single dose of one milligram of dexamethasone sodium phosphate
2. Patient is currently implanted with a pacemaker, ICD, or CRT-D/P device
3. Patient has had a previous unsuccessful attempt to place a lead in the LBB area
4. Patient has planned cardiac surgical procedures or interventional measures within 3 months after implant
5. Patient is expected to receive a heart transplant within 6 months
6. Patient life expectancy less than 6 months
7. Patient has the presence of another life-threatening, underlying illness separate from their cardiac disorder
8. Patient is enrolled or planning to enroll in another clinical trial that might confound the results of the present study
9. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
10. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Infection Rate | 0-6 months
  Rate of Infection
Perforation Rate | 0-6 months
  Perforation includes cardiac perforation, septal perforation, coronary sinus dissection, pericardial effusion, and cardiac tamponade.
Malfunction Rate | 0-6 months
  Malfunction includes 1) mechanical lead failure including lead insulation issues, lead fracture, and other lead damage, dysfunction, helix damage or fracture; malfunction or failure; and 2) electrical abnormalities of unknown cause including sensing issues, pacing issues, loss of capture, impedance abnormality, and noise; 3) excludes infection, perforation or dislodgement caused inappropriate therapy.
Cardiovascular Injury Rate | 0-6 months
  Cardiovascular Injury is a safety measure specific to LBBAP leads and includes Acute coronary syndrome; Coronary artery fistula; Coronary vein fistula/injury and Septal hematoma. This parameter also includes the right bundle branch block and complete heart block (permanent).
Implant success rate | At the time of implant
  Rate of Implant success of LBBAP lead
Lead dislodgement rate | 0-6 months
  Rate of LBBAP lead dislodgement
Pacing threshold | 0-6 months
  Measure of minimum electrical energy required to stimulate and depolarize
Impedence | 0-6 months
  Measure of lead impedance
Sensing Amplitude | 0-6 months
  Measure of lead sensing amplitude

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Fortis Escorts Heart Institute, New Delhi, National Capital Territory of Delhi
  - Meenakshi Mission Hospital & Research Centre, Madurai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No